CLINICAL TRIAL: NCT01755130
Title: Multimode Laser Optoacoustic Ultrasonic Tomography System for Breast Cancer Care
Brief Title: Laser Optoacoustic and Ultrasonic Imaging System Assembly in Finding Changes in Tumors in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to lack of funding
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-0210; NCI-2014-01243 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2013-00149; 2012-0210 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Breast Neoplasm; Inflammatory Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms

ARMS (1):
- Diagnostic (LOUISA 3D) (Experimental): Patients undergo LOUISA 3D over approximately 30 minutes on the same day or within 7 days of any breast imaging procedure and within 7 days before biopsy.
  Interventions: Procedure: Photoacoustic Imaging

INTERVENTIONS:
Procedure: Photoacoustic Imaging — Undergo LOUISA 3D

SUMMARY:
This clinical trial studies laser optoacoustic and ultrasonic imaging system assembly in finding changes in tumors in patients with breast cancer. Diagnostic procedures, such as laser optoacoustic and ultrasonic imaging system assembly, may help find and diagnose breast cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To successfully obtain images from laser optoacoustic and ultrasonic imaging system assembly (LOUISA) 3-dimensional (3D) and assess pathology in order to guide image calibration and gain knowledge about LOUISA 3D capabilities to detect and differentiate breast tumors.

II. Estimate and compare the false positive rate of LOUISA-3D compared to standard of care ultrasound for detecting breast cancer in year 5 of the study.

SECONDARY OBJECTIVES:

I. Determine optimal scanning parameters by assessing certain machine parameters (e.g. illumination and detection conditions, laser pulse repetition rate, laser ultrasound emission characteristics, type of imaging probe, two-dimensional images vs three-dimensional images, coupling medium characteristics, software and firmware, etc.), anatomical information (speed of sound image, acoustic attenuation image, acoustic scattering image), and functional information (total hemoglobin distribution [THb]/image of angiogenesis density, image of blood oxygen saturation [SO2], and image of water distribution).

OUTLINE:

Patients undergo LOUISA 3D over approximately 30 minutes on the same day or within 7 days of any breast imaging procedure and within 7 days before biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Mass palpable or nonpalpable
* Tissue density - all tissue types
* Menses - any stage of cycle
* Suspicious breast mass(es) defined by mammography or ultrasound indicating biopsy is needed (biopsy not needed if previous biopsy results are available on target lesion[s])
* Tumor location - the mammography or ultrasound report should not say that the tumor is in close proximity of chest wall
* Any tumor type (patients with inflammatory breast cancer may be included)

Exclusion Criteria:

* Patient is unable or unwilling to give informed consent for any reason
* Disability (psychiatric, neurological or physical, which precludes examination)
* Patient has tattoos on the region of interest
* Overweight over 250 pounds (LB)
* Very large breast size exceeding 6 inch diameter
* Patient has body piercing jewelry through the nipple that cannot be removed
* Patient has had a core or excisional biopsy in the ipsilateral breast within the last 2 weeks (patients with previous fine needle aspirations but no ultrasound evidence of hematoma or post biopsy [bx] change may be included)
* Patient has inflammatory skin disease (i.e., psoriasis, eczema) or other irritation affecting the breast
* Patient has any pain or high sensitivity in the breast
* Currently taking hormonal replacement therapy
* Non-ambulatory or unable to comply with exam
* Pregnant (pregnancy test is not required, only as confirmed by patient)
* Breastfeeding
* Prior breast treatment for target lesion
* Previous surgery of the breast in the last 3 months

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Number of images successfully obtained from laser optoacoustic and ultrasonic imaging system assembly (LOUISA) 3-dimensional (3D) | Within 7 days of the standard of care ultrasound
  Pathology will provide useful information including but not limited to type of malignancy, tissue type, and other qualitative information that is necessary for image calibration.
False positive rate of LOUISA 3D and standard of care ultrasound | Within 7 days of the standard of care ultrasound
  McNemar's test will be used to compare paired proportions and relative false positive rates.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org